CLINICAL TRIAL: NCT01782144
Title: Effect of Weight Loss on Foot Structure and Function in Obese Adults: A Pilot Study
Brief Title: Effects of Weight Loss on Foot Structure and Function in Obese Adults: A Pilot Study
Acronym: WLF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 12887
Record Dates: First submitted 2013-01-30; First posted 2013-02-01 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Obesity
Keywords: Obesity; Foot pain
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NutriSystem (Active Comparator): weekly behavior group weight loss education
  Interventions: Other: NutriSystem portion-controlled pre-packaged meals
- Education (Placebo Comparator): monthly behavior group weight loss education
  Interventions: Other: NutriSystem portion-controlled pre-packaged meals

INTERVENTIONS:
Other: NutriSystem portion-controlled pre-packaged meals

SUMMARY:
Obesity is a serious medical, social, and economic problem and is becoming even greater concern, as the prevalence of overweight and obese individuals has steadily increased over the years. Excessive body weight can have a profound influence on lower extremities, including pain, degenerative disease, and compromised quality of life. However, no study to-date has examined the effects of weight change on foot structure and function in individuals over time. The purpose of this study is to determine the effects of weight reduction on foot structure and function in obese adults. Improved understanding of the relationship between body weight and foot biomechanics is needed to promote health and healthier lifestyles.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 50 to 75, inclusive
* Body Mass Index is ≥ 30 kg/m2 but < 45 kg/m2 and body weight < 300 pounds
* Able to ambulate safely without the use of a walking aid (cane, crutches, or walker)
* Able to understand the information in the informed consent form and is willing and able to comply with the study-related procedures

Exclusion Criteria:

* Diabetes, stroke, end stage kidney disease requiring hemodialysis, or widespread malignant disease, gallbladder disease
* Severe peripheral vascular disease (defined as 1 < palpable pedal pulse and claudication pain in less than two blocks)
* Pregnant or nursing, as weight and hormonal changes during pregnancy may affect foot structure and function, which could confound the results of the study. Therefore, women who are pregnant or nursing will be excluded from the study.
* Not willing or able to make the required quarterly follow-up visits
* Insufficient (corrected) vision to complete the questionnaires
* Food allergies to the Nutrisystem, Inc. meal plan used in this protocol
* Participation in another formal weight loss program within last 6 months
* Uncontrolled hypertension (systolic blood pressure > 180 or diastolic blood pressure > 100 mmHg). Participants on medication treating hypertension for at least three months are allowable.
* Known atherosclerotic cardiovascular disease
* History of congestive heart failure
* History of a non-skin malignancy within the previous 5 years
* Any major active rheumatologic, pulmonary, hepatic, renal, dermatologic disease or inflammatory condition

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Walking speed | 3 months
  Change in walking speed at 3 month
Postural stability | 3 months
  Change in Fall Risk Test Score as measured by the BioDex Balance System.
Peak plantar pressure | 3 months
  Change in dynamic peak plantar pressure during barefoot walking.
Instruments of pain and disability | 3 months
  Change in answers on the following questionnaires: Revised Foot Function Index, the Medical Outcomes Study Short Form 36 (SF-36), Western Ontario and McMaster Universities Osteoarthritis Index.

SECONDARY OUTCOMES:
Arch Height Drop | 3 months
  Change in arch height in standing compared to sitting
Activities of Daily Living | 3 months
  Change in 50' walk time and pain, stair ascend/descend time and pain, and sit-to-stand.

CONTACTS AND LOCATIONS:
Overall Officials: Jinsup Song, DPM, PhD, Principal Investigator — Temple University
Locations (1):
- Gait Study Center, Philadelphia, Pennsylvania, United States